CLINICAL TRIAL: NCT04170400
Title: Observational Study Comparing Thin Pvc With Thick Silicone Gastric Calibration Tube for Bariatric Surgery
Brief Title: Observational Study Comparing Gastric Calibration Tubes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, Prof Dr, AZ Sint-Jan AV
Other Study IDs: 2019OSgastrictube
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study comparing thin pvc with thick silicone gastric calibration tube for bariatric surgery.

Most of the times a thin gastric tube is used. Sometimes insertion is difficult due to kinking, resistance, bulging and not advancing in the right spot requiring re introduction, help from a colleague, or change to the thick silicone type. When tube is changed during insertion to the silicone type the method insertion is compared with the previous approach.

DETAILED DESCRIPTION:
Observational study comparing thin pvc with thick silicone gastric calibration tube for bariatric surgery.

Most of the times a thin gastric tube is used. Sometimes insertion is difficult due to kinking, resistance, bulging and not advancing in the right spot requiring re introduction, help from a colleague, or change to the thick silicone type. When tube is changed during insertion to the silicone type the method insertion is compared with the previous approach.

A note is made of the problem encountered, how long it took to place it correctly ( time from insertion till first staple), what was done to solve the problem, if a new identical tube was used or another and what type was used. If another tube how log did it take to get first stapler done.

some demographic and procedure information is recorded: gender, age, BMI, procedure planned, first bariatric procedure or second after ...

ELIGIBILITY:
Inclusion Criteria:

* bariatric surgery being sleeve gastrectomy, gastric bypass or conversion procedure.

Exclusion Criteria:

* pre existing esophageal disease making use of gastric tube contra indicated, difficult or impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient sheduled for bariatric surgery > 18 year sold and most of the time morbid obese. BMI > 35
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
need to change gastric tube | intraoperative
  rate of changing gastric tube
introduction time | intraoperative
  time from start insertion till first staple in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Mulier, Principal Investigator — AZ Sint-Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium